CLINICAL TRIAL: NCT05787405
Title: CORONABED.BOT: an Automation Project Using Artificial Intelligence for Early Diagnosis of Clinical Evolution From SARS-CoV-2"
Brief Title: Early Diagnosis of Clinical Evolution From SARS-CoV-2
Acronym: CORONABEDBOT
Status: Completed | Type: Observational
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Responsible Party: Sponsor
Other Study IDs: CORONABED.BOT-COVID19- 3447
Record Dates: First submitted 2023-03-16; First posted 2023-03-28 (Actual); Last update posted 2025-03-12 (Actual); Status verified 2025-03

CONDITIONS: SARS-CoV-1 Infection
MeSH Terms: conditions — Severe Acute Respiratory Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Artificial Intelligence methods — The aim of the CORONA.BOT project is to exploit the Artificial Intelligence methods of Generator Real World Data Facility to automatically extract structured and unstructured data from hospital databases and to implement an early risk assessment (warning system) regarding the negative outcome for patients infected with SARS-CoV-2.

SUMMARY:
The aim of the CORONA.BOT project is to exploit the Artificial Intelligence methods of Generator Real World Data Facility to automatically extract structured and unstructured data from hospital databases and to implement an early risk assessment (warning system) regarding the negative outcome for patients infected with SARS-CoV-2.

The objective of CORONABED.BOT is to analyze the care pathways of patients from the same cohort as CORONA.BOT, in order to identify the total length of stay, intensive care occupations and flows between departments, based on variables demographics and first entry clinics Early identification of patients with symptoms compatible with SARS-CoV-2 infection will enable more rapid activation of isolation procedures, contact monitoring/contact history and decisions on the most appropriate clinical pathway in terms of type of treatment and unit. Similarly, the identification of factors correlated with worse outcomes will allow more effective planning for the use of critical resources (such as intensive care and others).

ELIGIBILITY:
Inclusion Criteria:

* adult patients (18 years of age or older)
* admitted to the Gemelli and Columbus Polyclinic
* diagnosis of SARS-CoV-2 infection (suspected cases will also be included).

Exclusion Criteria:

* aaaa

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: adult patients
Sampling Method: Probability Sample
Enrollment: 8000 (Actual)
Dates: Start 2020-12-01 (Actual); Primary Completion 2023-06-15 (Actual); Study Completion 2024-01-10 (Actual)

PRIMARY OUTCOMES:
the implementation of prediction models | 24 months
  tThe DataMart built will allow the creation of predictive models both for diagnosis of SARS-coV-2 pneumonia as well as death

CONTACTS AND LOCATIONS:
Overall Officials: Rita Murri, Principal Investigator — Fondazione Policlinico Universitario A. Gemelli, IRCCS
Locations (1):
- Fondazione Policlinico Gemelli, Rome, Italy

IPD SHARING:
Plan to Share IPD: No